# Cover Page for Informed Consent Document

Official Study Title: What makes people better at retrieving difficult words?

NCT05066750

Document Date: 1/3/22

 Version Date: 1.16.2019

Protocol Number: 2020-005



# University of Colorado Colorado Springs (UCCS) Consent to be a Research Subject

**Title:** What makes people better at retrieving difficult words?

**Principal Investigator**: Lori James, PhD

**Funding Source**: National Institutes of Health

**Key Information** You are being asked to choose whether or not you would like to participate in a research study. This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to produce words in response to definitions. You will watch a video, then see definitions and try to come up with a word that fits each one. You will also complete some surveys and other measures. Participation will take approximately 60 - 75 minutes. There are minimal risks involved in this study, but you may feel frustrated by the difficulty of the word production task or you might become bored with the surveys. Collected data will be stored by an identification code, not your name. You will not directly benefit from this study, but it will give researchers a better understanding of how individuals' personality and cognitive traits and setting in which naming occurs correspond with their ability to produce individual words.

#### Introduction

You are being asked to be in a research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study.

Before making your decision:

- Please carefully read this form or have it read to you.
- Please ask questions about anything that is not clear.

Feel free to take your time thinking about whether you would like to participate. By agreeing to be in the study you will not give up any legal rights. You may want to print a copy of the consent form for your records.

<u>Study Overview</u> This study is being conducted to learn more about how various personal and situational factors relate to the ability to produce difficult words that fit definitions. Results will be presented as group averages, not as individual responses. Your de-identified data may be made publicly available in a repository but will not be able to be connected to you. Findings may be published in journal articles and presented at conferences.

<u>Procedures</u> You are being asked to be in this research study because you are 18-30 or 65-80 years of age and a native, fluent speaker of American English. If you choose to participate, you will engage in a videoconference call with a researcher and also complete some surveys on Qualtrics. You will first complete a questionnaire about your personal information and then watch a brief video, following which you will be asked to provide words to fit definitions. We will record the word production task for later scoring. You will then take a vocabulary test and complete a few surveys. People over age 65 will complete one additional set of cognitive questions at the end of the study. The entire procedure will take approximately 60 – 75 minutes to complete.

Other people in this study: Approximately 200 people will participate in this study.

 Version Date: 1.16.2019

<u>Risks and Discomforts</u> There is minimal risk involved in this study. You might feel frustrated by the word production task, or you might become bored while completing the surveys. This discomfort is not expected to be greater than that experienced during everyday life. You may stop participating in the study at any time without any negative consequences.

<u>Benefits</u> You will not directly benefit from this study, but it will give researchers a better understanding of how individuals' personal traits and situational factors relate to the ability to produce difficult words.

<u>Compensation</u> UCCS student participants are compensated with 2.5 SONA system credits. Non-student participants are compensated with a \$12 electronic gift card.

<u>Confidentiality</u> None of your data will have your name attached to it, nor will the recording. Participant information will be kept separately from data, in a secure location. Participant information and data will be stored only by a meaningless participant identification code. Only Dr. James and her research assistants will have access to raw or coded data. All electronic data files will be kept on password-protected computers.

Certain offices and people other than the researchers may have access to study records. Government agencies and UCCS employees overseeing proper study conduct may look at your study records. These offices include the UCCS Institutional Review Board, and the UCCS Office of Sponsored Programs and Research Integrity. UCCS will keep any research records confidential to the extent allowed by law. A study number rather than your name will be used on study records wherever possible. Study records may be subject to disclosure pursuant to a court order, subpoena, law or regulation.

## Voluntary Participation and Withdrawal from the Study

Taking part in this study is voluntary. You have the right to leave the study at any time without penalty. You may refuse to answer any questions that you do not wish to answer. If you withdraw from the study, you may request that your data not be used by contacting the Principal Investigator listed above and below. If you are a UCCS student, there are alternative options to earn credit other than participating in this study. Contact your course instructor if you would like to learn about alternatives for receiving extra credit.

This trial will be registered and may report results on www.ClinicalTrials.gov.

### **Contact Information**

Protocol Number: 2020-005

Contact (PI's info): Lori James at ljames@uccs.edu

- if you have any questions about this study or your part in it,
- if you have questions, concerns or complaints about the research, or
- if you would like information about the survey results when they are prepared.

Contact the Research Integrity Compliance Program Director at 719-255-3903 or via email at irb@uccs.edu:

- if you have questions about your rights as a research participant, or
- if you have questions, concerns or complaints about the research.

#### **Electronic Consent**

Please print a copy of this consent form for your records, if you so desire.

I have read and understand the above consent form, I certify that I am 18 years old or older and, by clicking the button to enter the survey, I indicate my willingness to voluntarily take part in the study.

 Version Date: 1.16.2019